CLINICAL TRIAL: NCT06716008
Title: Effect of Manual Diaphragmatic Release on Ventilatory Functions in Women With Rheumatoid Arthritis
Brief Title: Manual Diaphragmatic Release on Ventilatory Functions in Women With Rheumatoid Arthritis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Middle East University (Other)
Responsible Party: Principal Investigator, Saher Lotfy El Gayar, Assistant Professor of Physical Therapy, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Manual Diaphragmatic Release
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Rheumatic Arthritis; Lung Function
MeSH Terms: conditions — Rheumatic Fever

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual diaphragmatic release group (Active Comparator): 30 women with rheumatoid arthritis who will receive low to moderate intensity aerobic training plus manual diaphragmatic release
  Interventions: Other: Aerobic training; Other: Manual Diaphragm Release
- Control group (Active Comparator): 30 women with rheumatoid arthritis who will receive low to moderate intensity aerobic training only.
  Interventions: Other: Aerobic training

INTERVENTIONS:
Other: Aerobic training — For twelve weeks, the women in the study group will participate in aerobic training on cycle ergometer. Each session will consist of 30-45 minutes of cycling at a moderate intensity, accompanied by a workout heart rate ranging from 65% to 75% of the maximal heart rate and ranging between 12 and 14 on the Borg rating of perceived exertion 20-point scale. After ten minutes of warm-up, every session will end with a brief 3-minute period of cool-down.
Other: Manual Diaphragm Release — The participant will assume a supine position with relaxed limbs. The therapist should position themselves at the head of the participant and make manual contact with the pisiform, hypothenar region, and the last three fingers on both sides, underneath the seventh to tenth rib costal cartilages. The therapist's forearms should be aligned towards the participant's shoulders. During the inspiratory phase, the therapist gently pulled the points of contact with both hands in the direction of the head and slightly laterally, accompanying the elevation of the ribs. Therapist progressively increases the depth of their contact within the costal margin.
  Arms: Manual diaphragmatic release group

SUMMARY:
Evaluate the effect of manual diaphragmatic release on ventilatory functions in women with rheumatoid arthritis

DETAILED DESCRIPTION:
Sixty women with rheumatoid arthritis will be sourced from the rheumatology outpatient clinic at Tanta University hospitals in Egypt, with referrals from rheumatologists. Patients will be randomly assigned into two groups.

The study group will include 30 women participating in manual diaphragmatic release plus aerobic training for 12 weeks while the control group will include 30 women participating in aerobic training only for 12 weeks. At baseline and poststudy, the following outcomes will be assessed:

1. Ventilatory functions (Forced vital capacity and total lung capacity).
2. Functional capacity using modified Bruce treadmill incremental exercise test (Maximal oxygen consumption estimation).
3. Quality of life (Short form health survey).

ELIGIBILITY:
Inclusion Criteria:

* All women will have rheumatoid arthritis for more than 2 years with low-to-moderate disease activity.
* Normal to mildly restrictive lung pattern.
* Their ages will be ranged from 40 to 60 years old.
* Their body mass index will be less than 30 Kg/m2.

Exclusion Criteria:

* Chronic chest diseases.
* Recent parenteral steroid administration.
* Cardiovascular disorders (coronary heart disease, heart failure, cardiac arrhythmia, peripheral arterial disease, uncontrolled hypertension).
* Smokers.
* Joint surgery (in the preceding 6 months).
* Musculoskeletal/ neurological limitations to exercise.
* Pregnancy.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Females
Enrollment: 60 (Estimated)
Dates: Start 2024-12-03 (Estimated); Primary Completion 2025-03-10 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Ventilatory function | At baseline and 12 weeks
  Ventilatory function parameters, including forced vital capacity and forced expiratory volume in the first second will be measured by experienced technicians at baseline and after 12 weeks in all groups using the Medgraphics pulmonary function testing system (Breezesuite Ultima PFX, Milano, Italy) in strict adherence to the guidelines outlined in the user manual.

SECONDARY OUTCOMES:
Functional capacity | At baseline and after 12 weeks
  Cardiopulmonary exercise test will be conducted for all women at baseline and post-study based on the guidelines set by the American College of Sports Medicine to determine maximal oxygen consumption for each women.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Sayed Saif, Ph.D, Study Director — National institute for Gerontology

IPD SHARING:
Plan to Share IPD: No